CLINICAL TRIAL: NCT02028598
Title: A Randomized, Open-labeled, 6-sequence, 3-period, 3-treatment Crossover Study to Evaluate the Effect of Co-administration of Clomipramine HCl (Condencia Tab.) 15mg and Sildenafil Citrate (Viagra Tab.) 100mg on the Safety and Pharmacokinetic/Pharmacodynamic Properties of Clomipramine and Sildenafil Compared to the Effects After Single Oral Administration in Healthy Male Volunteers
Brief Title: Drug-Drug Interaction of Clomipramine HCl and Sildenafil Citrate in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTC Bio, Inc. (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTC-PED-DDI-1
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Clomipramine; Premature ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Clomipramine; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence A (Experimental): Treatment 1 - Treatment 2 - Treatment 3
  Interventions: Drug: Treatment 1; Drug: Treatment 2; Drug: Treatment 3
- Sequence B (Experimental): Treatment 1 - Treatment 3 - Treatment 2
  Interventions: Drug: Treatment 1; Drug: Treatment 2; Drug: Treatment 3
- Sequence C (Experimental): Treatment 2 - Treatment 1 - Treatment 3
  Interventions: Drug: Treatment 1; Drug: Treatment 2; Drug: Treatment 3
- Sequence D (Experimental): Treatment 2 - Treatment 3 - Treatment 1
  Interventions: Drug: Treatment 1; Drug: Treatment 2; Drug: Treatment 3
- Sequence E (Experimental): Treatment 3 - Treatment 1 - Treatment 2
  Interventions: Drug: Treatment 1; Drug: Treatment 2; Drug: Treatment 3
- Sequence F (Experimental): Treatment 3 - Treatment 2 - Treatment 1
  Interventions: Drug: Treatment 1; Drug: Treatment 2; Drug: Treatment 3

INTERVENTIONS:
Drug: Treatment 1 — An oral single dose administration
  Other Names: Clomipramine HCl 15mg (Condencia Tab)
Drug: Treatment 2 — An oral single dose administration
  Other Names: Sildenafil citrate 100mg (Viagra Tab)
Drug: Treatment 3 — Co-administration of oral single doses
  Other Names: Clomipramine HCl 15mg (Condencia Tab); Sildenafil citrate 100mg (Viagra Tab)

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics/pharmacodynamics of co-administration of Clomipramine HCl 15mg and Sildenafil citrate 100mg compared to the effects after single oral administration in Korean healthy male volunteers.

DETAILED DESCRIPTION:
Clomipramine is a dibenzazepine-derivative tricyclic antidepressant (TCA) and is a potent inhibitor of serotonin and norepinephrine reuptake. Clomipramine may be used in a variety of indications. Condencia Tab contains low dose of 15mg of clomipramine HCl as an active ingredient, which is newly approved to market for the treatment of premature ejaculation.

This study is a prospective, randomised, open-labeled, 6-sequence, 3-period, 3-treatment, crossover, and single-center clinical trial. A total of 30 healthy male volunteers will be enrolled and randomised into one among 6 groups (5 subjects per a group). The safety and PK/PD characteristics of co-administration of Clomipramine HCl and Sildenafil citrate will be investigated closely compared to the effects after single dose administrations.

ELIGIBILITY:
Inclusion Criteria:

* Korean healthy males aged between 19 and 65
* Body weight between 60kg and 90kg, BMI between 19 and 27
* Given informed consent

Exclusion Criteria:

* Clinically significant medical history and/or concurrent disease
* SBP >=140 mmHg or <=90 mmHg, DBP >=95 mmHg or <=50 mmHg
* Orthostatic hypotension
* Hypersensitivity to any ingredient of investigational drugs
* Severe bleeding or blood donation within 8 weeks prior to study participation
* Alcoholism or drug abuser
* Smoking more than 0.5 pack-year
* Persistent alcohol consumption more than 21 units(210g)/week
* Participation in other investigational clinical trial

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The systemic exposure measured as area under the curve (AUC) | From Day 1(dosing) to Day 4(72hrs)
The maximum concentration (Cmax) | From Day 1(dosing) to Day 4(72hrs)

SECONDARY OUTCOMES:
Pharmacokinetic parameters except the primary endpoints | From Day 1(dosng) to Day 4(72hrs)
  Including Tmax, T1/2, AUCnorm, Cmax norm, CL/f and Cmax/AUC
The maximum change of systolic blood pressures within 12hrs after dosing | Day 1(dosing) to Day 2(12hrs)
  At supine and upright positions
Adverse events | For 3 Weeks after dosing
The maximum change of dystolic blood pressure within 12hrs after dosing | From Day 1(dosing) to Day 2(12hrs)
  at supine and upright positions
The maximum change of heart rates within 12 hours after dosing | From Day 1(dosing) to Day 2(12hrs)
  At supine and upright positions
The rate of the subjects who experienced the clinically significant change of blood pressures | From Day 1(dosing) to Days 2(12hrs)
  Clinically significant changes will be classified into 4 groups: SBP change >=30 or 20 mmHg, DBP change >= 20 or 10 mmHg (at supine and upright positions)

CONTACTS AND LOCATIONS:
Overall Officials: Yun Hi Kang, M.D., Principal Investigator — Yangji Hospital
Locations (1):
- Yangji Hospital, Seoul, South Korea